CLINICAL TRIAL: NCT06877858
Title: A Dose-Finding Study of Methadone Loading Dose Initiation for Opioid Use Disorder With Fentanyl Use
Brief Title: MethaLoad Dose-Finding Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ashish P Thakrar, MD MS, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 857972
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder (OUD)
Keywords: methadone; fentanyl; opioid use disorder; opioid addiction; opiate addiction; OUD
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methadone

STUDY DESIGN:
Intervention Model Description: Bayesian Optimal Interval Design (BOIN) for dose-finding studies
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) (Active Comparator): Day 1: 40mg oral methadone Day 2: 40mg oral methadone
  Interventions: Drug: Methadone hydrochloride
- Loading Dose (Experimental): Day 1: loading dose (60mg, 80mg, 100mg, or 120mg oral methadone) Day 2: 50% of the loading dose (30mg, 40mg, 50, or 60mg oral methadone)
  Interventions: Drug: Methadone hydrochloride

INTERVENTIONS:
Drug: Methadone hydrochloride — Methadone loading dose initiation (vs. standard initiation in the TAU arm)

SUMMARY:
The goal of this study is to develop a loading dose approach to starting methadone to treat opioid use disorder with fentanyl use ("fentanyl OUD", herein). This study is a participant- and assessor- blinded dose-finding study using the Bayesian optimal interval (BOIN) design. Investigators aim to recruit n=24 participants with fentanyl OUD to a research unit for monitored methadone initiation. Participants will be randomized to standard initiation vs. loading dose initiation at one of four doses.

ELIGIBILITY:
Inclusion criteria:

1. Male, female, transgender, or non-binary, aged 18 years or older
2. DSM-5 criteria for opioid use disorder, moderate-severe
3. Fentanyl positive urine drug test
4. Able to provide a dated & written informed consent in English prior to the conduct of any study related procedures
5. Stated willingness to comply with all study procedures and availability for the duration of the study
6. Ability to take oral medication and be willing to adhere to the dosage regimen
7. Interest in starting methadone treatment for opioid use disorder at one of three locations: Merakey Parkside at 5000 Parkside, Merakey 5429 Germantown Avenue, or Merakey 1745 North 4th Street
8. Reliable access to a working phone

Exclusion criteria:

1. Hypersensitivity or allergy to methadone that is previously documented
2. Pregnancy or actively lactating (with urine pregnancy test performed on screening and repeated on admission to the unit prior to randomization)
3. Taking medications for opioid use disorder, per self-report or per urine drug testing detection of buprenorphine or methadone
4. At risk of benzodiazepine or alcohol withdrawal as defined by: prior benzodiazepine or alcohol withdrawal in the past 3 months, current daily use of benzodiazepines or alcohol, or DSM-5 criteria for hypnotic-sedative or alcohol use disorder
5. At risk of severe medetomidine withdrawal based on: serum or urine testing for medetomidine (if available), prior withdrawal syndrome requiring intensive care unit admission within past 6 months, and/or severe nausea/vomiting during first 4 hours of withdrawal, at the discretion of the study physicians
6. At risk for methadone-induced QT-prolongation: prolonged QTc on screening or admission EKG (greater than 450ms in men, greater than 460ms in women), history of QT prolongation, previously documented long QT syndrome, history of ventricular arrhythmia (e.g., torsades de pointes), history of cardiac hypertrophy, history of cardiac conduction abnormalities, taking medications that affect cardiac conduction (at study physician discretion; including but not limited to: amiodarone, flecainide, sotalol, azithromycin, ciprofloxacin, levofloxacin, citalopram, escitalopram, hydroxychloroquine, chlorpromazine, haloperidol, donepezil, ibogaine, cilostazol), serum potassium concentration less than 3.5 mg/dL, or serum magnesium concentration less than 1.7 mg/dL.
7. Significant hepatic dysfunction, defined as: AST and/or ALT 3x upper limit of normal, or total bilirubin 1.5x upper limit of normal
8. Significant renal dysfunction, defined as: eGFR less than or equal to 60 mL/min
9. Chronic hypotension (<90/50 mmHg) or episodic symptomatic hypotension, defined as a history of active or recurrent orthostatic hypotension or syncope
10. Significant pulmonary disease, defined as: baseline SpO2 <95% on screening or admission, requiring oxygen at home (chronically or at bedtime), or COPD with modified MRC Dyspnea Scale greater than 2 ("I stop for breath after walking about one city block")
11. Suspected gastrointestinal obstruction, per medical history
12. Active, chronic use of the CYP3A4-inducers or -inhibitors rifampin, phenytoin, St John's wort, phenobarbital, carbamazepine, voriconazole, efavirenz, nelfinavir, nevirapine, ritonavir, and lopinavir/ritonavir, abacavir, or amprenavir
13. Pending legal action that could prohibit participation and/or compliance in study procedures
14. Presence of any other psychiatric and/or medical disorder that, in the opinion of the PI, will interfere with completion of the study or place the patient at heightened risk through participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rate | 24 hours
  The primary objective of the study is to identify a methadone loading dose approach appropriate for future study as an alternative initiation strategy for individuals with OUD using fentanyl or other high-potency synthetic opioids.
  The loading dose appropriate for future study will be identified as the highest loading dose with a dose-limiting toxicity (DLT) rate less than 10%. DLT definition: the proportion of individuals in each loading dose arm who meet any one of four safety outcomes within 24 hours of methadone loading dose administration: (1) Richmond Agitation-Sedation Scale (RASS) less than -1, (2) respiratory rate (RR) less than 8 breaths per minute, (3) peripheral oxygen saturation (SpO2) less than 92%, or (4) corrected QT interval (QTc) greater than 500ms.

SECONDARY OUTCOMES:
Opioid withdrawal severity | 24 hours
  Peak and time-weighted mean subjective opioid withdrawal (using the Subjective Opioid Withdrawal Scale, SOWS) and the Clinical Opiate Withdrawal Scale (COWS) over 24 hours after initial methadone dose
Opioid craving | 24 hours after initial methadone dose
  Peak and time-weighted mean opioid craving, using a visual analogue scale (VAS) assessment (1-100) over 24 hours after initial methadone dose
Peak plasma methadone concentration | 48 hours
  Peak plasma methadone concentration after initial loading dose (Day 1) and after first maintenance dose (Day 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Center for Studies of Addiction (CSA), Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol